CLINICAL TRIAL: NCT01171274
Title: Randomisierte Kontrollierte Studie Zum Einfluss Von Hatha Yoga Auf Sensorische Schwellen, Kinästhetik Und Körperbild Bei Patienten Mit Chronischen Nackenschmerzen
Brief Title: Effects of Hatha Yoga on Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Gustav J Dobos, MD, Universität Duisburg Essen, Chair of Complementary and Integrative Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-4358
Record Dates: First submitted 2010-07-23; First posted 2010-07-28 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Neck Pain
Keywords: neck pain; yoga; proprioception; sensory thresholds; randomized controlled trial
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hatha Yoga (Active Comparator): * 9 weeks of Hatha Yoga, designed for treating chronic neck pain, as a group intervention.
  * One class of 90 minutes per week, 10 minutes training at home each day.
  Interventions: Behavioral: Hatha Yoga
- Exercise information (Active Comparator): * 9 weeks of exercises practiced at home.
  * Patients receive detailed information regarding appropriate exercises and behaviour for chronic neck pain patients.
  Interventions: Behavioral: Information regarding exercises and behaviour

INTERVENTIONS:
Behavioral: Hatha Yoga — * 9 weeks of Hatha Yoga, designed for treating chronic neck pain, as a group intervention.
  * One class of 90 minutes per week, 10 minutes training at home each day.
  Arms: Hatha Yoga
Behavioral: Information regarding exercises and behaviour — * 9 weeks of exercises practiced at home.
  * Patients receive detailed information regarding appropriate exercises and behaviour for chronic neck pain patients.
  Arms: Exercise information

SUMMARY:
Hatha Yoga is a traditional system of exercises, used in India for the relief of painful condition since centuries and gaining more and more interest in Europe and the US. While studies have demonstrated benefits of Hatha Yoga for patients with chronic low back pain, no studies regarding chronic neck pain are available until now. The purpose of this study is to determine if Hatha Yoga can ameliorate chronic neck pain and related restrictions.

DETAILED DESCRIPTION:
Hatha Yoga is a traditional system of exercises, used in India for the relief of painful condition since centuries and gaining more and more interest in Europe and the US. The efficacy of Hatha Yoga for relieving chronic low back pain has been repeatedly demonstrated in clinical trials, while there are no studies in the literature regarding chronic neck pain. The aim of this study is to investigate, whether a 9 weeks-course of Hatha Yoga reduces subjective pain ratings and disability in patients suffering from chronic neck pain. Furthermore, as neck pain patients have been shown to suffer from impaired sensory processing and proprioception, along with restricted range of motion, the study aims to test if Hatha Yoga can improve these variables. Therefore, tests regarding cervicocephalic proprioception, active range of motion and the processing of mechanical, vibration and pain stimuli will be included.

58 patients with chronic nonspecific neck pain will be randomized to either Hatha Yoga group or control group, receiving information regarding exercises for chronic neck pain. The control group will be offered to take part in a Yoga class after the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Chronic mechanical neck pain, at least 40 mm on the 100mm visual analog scale.
* Pain for at least 3 months.

Exclusion Criteria:

* radicular symptoms
* congenital spine deformity
* pregnancy
* rheumatic diseases
* oncologic diseases
* other severe psychiatric or somatic comorbidity
* recent invasive or surgical treatment of the spine
* regularly yoga practice participation in other studies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Neck pain intensity (100mm visual analog scale) | Week 10
  100mm visual analog scale

SECONDARY OUTCOMES:
Cervicocephalic kinesthetic sensibility | Week 10
  The ability to exactly relocate the head on the trunk in a self-chosen "neutral" forward-position after an active movement.
  according to: Revel M, Andre-Deshays C, Minguet M. Cervicocephalic kinesthetic sensibility in patients with cervical pain. Arch Phys Med Rehabil. 1991;72:288-91.
Active range of motion | Week 10
  6 movement directions (flexion, extension, rotation right/left, lateral flexion right/left)
Pain related to motion | Week 10
  100mm visual analog scale for 6 movement directions (flexion, extension, rotation right/left, lateral flexion right/left)
  according to: Irnich D, Behrens N, Molzen H, König A, Gleditsch J, Krauss M, Natalis M, Senn E, Beyer A, Schöps P. Randomised trial of acupuncture compared with conventional massage and "sham" laser acupuncture for treatment of chronic neck pain. BMJ. 2001 Jun 30;322(7302):1574-8.
Pressure pain threshold | Week 10
  Pressure pain threshold measured at two individual points at the neck: (1) at the point of maximal pain and (2) in the adjacent region, one to two cm outside the painful area. Furthermore, it is measured bilaterally at levator scapulae muscle, semispinalis capitis muscle and trapezius muscle and at both hands, serving as control sites.
  Measurement procedure according to the protocol of QST. Reference: Rolke R et al.. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values. Pain 2006;123:231-243.
Neck disability index (NDI) | Week 10
  The Neck Disability Index is an instrument to assess neck pain complaints. Reference: Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther 1991;14:409-415.
SF-36 | Week 10
  The SF-36 is a short-form health survey consisting of 8 scales (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, mental health) measuring functional health and well-being as well as a physical a and mental health component scores.
  Reference: Bullinger M, Kirchberger I. SF-36 Fragebogen zum Gesundheitszustand. Göttingen: Hogrefe, 1998.
Pain diary | From Week 1 to Week 10
  100mm visual analog scale for rating neck pain intensity each day

CONTACTS AND LOCATIONS:
Locations (1):
- Kliniken Essen-Mitte, Knappschafts-Krankenhaus, Department for Internal and Integrative Medicine, Essen, North Rhine-Westphalia, Germany